CLINICAL TRIAL: NCT05882461
Title: 90Second Caregiver: A Randomized Control Trial of an E-health Letter for Caregivers
Brief Title: An E-health Letter Intervention for Caregivers
Acronym: 90Second
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1025834
Record Dates: First submitted 2021-03-15; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Caregivers; Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a two-arm Randomized Control Trial (RCT), comparing a group assigned to receive the 90Second Caregiver Caregiver health letter, with a usual care control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In sequence of eligibility, participants will be randomized to the treatment arm or the control arm, with a 1:1 allocation ratio stratified by gender. The randomization sequence will be generated by a trained person that is not related to the study participants in any way. The investigators and study staff will be blinded to the randomization sequence until the end of the study. Participant randomization will be performed in REDCap. REDCap maintains an automated audit trail which includes the assigned study identification number, treatment allocation, and date and time of the allocation assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Those receiving the 90Second Caregiver health letter (Experimental): The 90Second Caregiver health letter is a weekly online publication that addresses topics relevant for caregivers. It combines scientifically-valid, evidence-based information with actionable tips to improve caregiver self efficacy and well-being. Participant in this group will receive a 90Second Caregiver health letter every week, via email.
  Interventions: Behavioral: 90Second Caregiver health letter
- The usual care control group (No Intervention): Participants that are randomized to be in the usual care control group will continue on as participants in the Caring Forward Trials within Cohort Study (i.e. filling out questionnaires every 6-months). Participants will continue to participate in the Caring Forward Study until completion in March 2022.

INTERVENTIONS:
Behavioral: 90Second Caregiver health letter — Participant receives the weekly health letter via email
  Arms: Those receiving the 90Second Caregiver health letter

SUMMARY:
The purpose of the present study is to conduct a two-arm Randomized Control Trial (RCT) comparing individuals receiving the 90Second Caregiver health letter, with a usual care (routine care received by caregivers) control group.

The goals of the present study are:

* To evaluate the effectiveness of the 90Second Caregiver health letter in improving caregiver's self-efficacy (primary outcome), savouring, and quality of life (secondary outcomes).
* To evaluate the effectiveness of the 90Second Caregiver health letter in reducing caregiver's psychological strain and caregiver burden (secondary outcomes).
* To examine the impact of levels of engagement with the 90Second Caregiver health letter on primary and secondary outcomes.
* To assess the usability of the 90Second Caregiver health letter, as it relates to the relevance of topic, user friendliness, and appropriateness of the readability levels.
* To evaluate psychometric properties of self-constructed measures in 90Second newsletter.

DETAILED DESCRIPTION:
The present study will examine the effectiveness of the 90Second Caregiver health letter in increasing self-efficacy in a sample of informal caregivers of ABI survivors in Nova Scotia. Participants in this study will be recruited from the Caring Forward Trials within Cohort Study (REB#1025253). The study is funded by the Nova Scotia Department of Health and Wellness.

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently enrolled in the Caring Forward Trials within Cohort study (REB#1025253)
* Participant has agreed to be contacted for future studies by Dr. McGrath's staff
* Participant has agreed for their data to be used for future studies
* Participant has mild levels of distress, as indicated by mild scores on the DASS-21 and/or the ZBI-SF

Exclusion Criteria:

* Participant is NOT currently enrolled in the Caring Forward Trials within Cohort study (REB#1025253)
* Participant has NOT agreed to be contacted for future studies by Dr. McGrath's staff
* Participant has NOT agreed for their data to be used in future studies
* Participant does NOT report mild levels of distress, as indicated by mild scores on the DASS-21 and/or the ZBI-SF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Caregiving self-efficacy | [Time Frame: At baseline.]
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | [Time Frame: Six months following baseline.]
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | [Time Frame: Twelve months following baseline.]
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | [Time Frame: Eighteen months following baseline.]
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | [Time Frame: Twenty four months following baseline.]
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.

SECONDARY OUTCOMES:
Psychological strain | [Time Frame: At baseline.]
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | [Time Frame: Six months following baseline.]
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | [Time Frame: Twelve months following baseline.]
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | [Time Frame: Eighteen months following baseline.]
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | [Time Frame: Twenty four months following baseline.]
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Caregiver burden | [Time Frame: At baseline.]
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | [Time Frame: Six months following baseline.]
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | [Time Frame: Twelve months following baseline.]
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | [Time Frame: Eighteen months following baseline.]
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | [Time Frame: Twenty four months following baseline.]
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Savouring | [Time Frame: At baseline.]
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | [Time Frame: Six months following baseline.]
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | [Time Frame: Twelve months following baseline.]
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | [Time Frame: Eighteen months following baseline.]
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | [Time Frame: Twenty four months following baseline.]
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Overall quality of life and general health | [Time Frame: At baseline.]
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | [Time Frame: Six months following baseline.]
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | [Time Frame: Twelve months following baseline.]
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | [Time Frame: Eighteen months following baseline.]
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | [Time Frame: Twenty four months following baseline.]
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.

OTHER OUTCOMES:
Usability of the 90Second Caregiver health letter | through study completion, an average of 1 year
  The current study will also assess the usability of the 90Second Caregiver health letter by evaluating the relevance of topic, learnability, and acceptability of the program. The usability questionnaire was developed for the current study.

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to indicate during Informed Consent whether their de-identified data may be shared with other researchers, provided the study is approved by an ethics board and researchers agree to use the data only for the purposes described in the approved research study. De-identified data from all outcome measures will be made available to approved researchers upon request, provided individual participants have provided consent.
Supporting Information: Study Protocol, SAP, ICF